CLINICAL TRIAL: NCT05615493
Title: The Effectiveness of Radial Extracorporeal Shock Wave Therapy as Additional Treatment Modality for Spastic Equinus Deformity in Chronic Hemiplegic Patients, A Double-Blinded, Randomized Controlled Study.
Brief Title: The Effectiveness of Radial Extracorporeal Shock Wave Therapy as Additional Treatment Modality for Spastic Equinus Deformity in Chronic Hemiplegic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Doaa Waseem Nada (Other)
Responsible Party: Sponsor-Investigator, Doaa Waseem Nada, Principal investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Tanta University35910
Record Dates: First submitted 2022-10-30; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Hemiplegic Patients
Keywords: Spasticity,; Equinus foot ,; Hemiplegia,; Extracorporeal shock wave
MeSH Terms: conditions — Muscle Spasticity; Hemiplegia

STUDY DESIGN:
Intervention Model Description: adult ischemic or hemorrhagic hemiplegic stroke patients with unilateral spastic equinus foot for at least 6 months before enrollment to reduce the confounding effect of natural recovery
Who Masked: Participant, Care Provider, Investigator
Masking Description: The closed envelop method will be used for the randomization of the patients who will be blinded to group allocation. The assessments will be done by the first physiatrist (A), who will not involved in patients' sessions. The randomization will be performed by the second physiatrist (B ) who will not be involved in patients' assessment and ESWT sessions . ESWT Sessions for both groups will be will be carried out by the third physiatrist (C ) who will not take part in the assessments or patients' randomization . Both (C) and (A) were blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Will receive rESWT once weekly for one month
  Interventions: Device: radial extracorporeal shock wave therapy
- Group II (Sham Comparator): Will receive Sham rESWT once weekly for one month
  Interventions: Device: sham radial extracorporeal shock wave therapy

INTERVENTIONS:
Device: radial extracorporeal shock wave therapy — Radial extracorporeal shock wave therapy (r ESWT) will be applied by Dornier AR2 machine (Dornier MedTech GmbH, Wessling, Germany) under ultrasound guidance, at musculotendinous junction of medial and lateral head of the gastrocnemius for spastic calf (gastrocnemius muscle and the soleus) muscles . 1.500 pulses will be applied by an R20 probe with a focusing depth of 4cm.The intensity will be 0.10 mJ to 0.3mJ/mm2 (2.5 bar), with frequency 4 Hz every week for one month .No anesthetic or analgesic drugs will be administered to patients during the therapy session
  Arms: Group I
Device: sham radial extracorporeal shock wave therapy — Dornier AR2 machine (Dornier MedTech GmbH, Wessling, Germany) used under ultrasound guidance, at musculotendinous junction of medial and lateral head of the gastrocnemius for spastic calf (gastrocnemius muscle and the soleus) muscles . 1.500 pulses will be applied by an R20 probe with intensity of 0.10 mJ to 0.3mJ/mm2 (2.5 bar), & frequency 4 Hz every week for one month without operating the machine .
  Arms: Group II

SUMMARY:
This is a prospective, double blinded randomized, placebo-controlled study that will be conducted on 112 adult ischemic or hemorrhagic hemiplegic stroke patients with calf muscles spasticity so as to evaluate the effectiveness of radial extracorporeal shock wave therapy (r ESWT) as an additional treatment modality for spastic equinus deformity in those patients. Allocation of patients into two groups after eligibility testing & randomization will be done:

Group I: patients will receive rESWT once weekly for one month , Group II: patients will receive Sham rESWT once weekly for one month. Each patient will be evaluated by the same well trained physiatrist for clinical, Electrophysiological and Musculoskeletal Ultrasound (MSKUS) assessments at baseline (t0), and after 1 month (t1) and after 2 months (t2) .

DETAILED DESCRIPTION:
Study design & Participants selection:

This is a prospective, randomized, placebo-controlled study that will be conducted from October 2022 to March 2023, on 112 consecutive adult ischemic or hemorrhagic hemiplegic stroke patients with calf muscles spasticity (grade 1 - 4) by the modified Ashworth scale (MAS) who will be recruited from out patient clinic of Rheumatology , Rehabilitation and Physical Medicine Department ,Tanta university Hospital, and will be assessed for study eligibility.

Inclusion criteria:

All patients who exhibited signs of unilateral spastic equinus foot for at least 6 months before the enrollment in the study will be selected to reduce the confounding effect of natural recovery.

Exclusion criteria:

Patients with fixed contractures or deformities at the ankle, fractures, cognitive impairment, different types of neuropathies or myopathies, implanted pacemaker and prior /or planned treatment using antispastic medications (i.e intrathecal baclofen or Botox injection ) or chemo -denervation ( phenol or alcohol nerve blocks ) within the last 6 months preceding the study , will be excluded.

Randomization :

The closed envelop randomization method will be used for the randomization of the patients who will be also blinded to group allocation.

The patients will be allocated into two groups after eligibility testing& randomization:

Group I: will be exposed to rESWT once weekly for one month Group II: will be exposed to Sham rESWT once weekly for one month. During the study period, oral anti-spastic medications and stretching exercises will be similarly given for both groups. Tizanidine hydrochloride will be the oral anti-spastic used at a daily dosage of 2 mg for first 4 days and then 4 mg until the end of the follow up period. Stretching exercises will be included and given at 30 min/day, at 5 weekly sessions over the treatment period. Stretching exercises as well as rESWT will be provided by the same blinded well-trained physiatrist and the patients in both groups will not be allowed to change the dose of anti-spastic medication during the study period.

The used assessment measures will be explained to all patients before having their written informed consents to participate in this study.

All data and results of the research will be used for scientific purposes with assurance of patient privacy.

Evaluation protocol and outcome measurements:

Each patient will be evaluated by the same well trained physiatrist for clinical, Electrophysiological and Musculoskeletal Ultrasound (MSKUS) assessments at baseline (t0), and after 1 month (t1) and after 2 months (t2) .

A. Clinical assessment :

1. Plantar-flexor muscles spasticity: will be assessed by modified Ashworth scale (MAS). It is a 5-point scale , ranging from ( 0 ) as normal muscle tone to (4 ) which is limb rigid in flexion or extension.
2. Passive ankle dorsiflexion motion (PADFM) : of the affected side will be measured with a goniometer while the patient is lying in a supine position with the knee flexed.. The readings will be recorded and the mean score will be calculated. The degree of ankle planter flexion will be measured as a negative value, and the degree of ankle dorsiflexion will be measured as a positive value.
3. The timed 10 meters walk test (10 MWT) :

The 10 Meter Walking Test (10 MWT) assesses short duration walking speed (m/s) & measures the time required to walk 10 meters. The time taken by the patients will be recorded by stopwatch ,two consecutive trials will be done and the mean time will be calculated .

B. Electrophysiological assessment:

The H/M ratio (Ratio of maximum H reflex to maximum M response), will be assessed using Electromyography machine (Neuroback ,Nihinon Kohden 4 channel. Japan 2008). The maximal amplitude of H-reflex will be obtained with low intensity, with gradual increase of the stimulus intensity, the M-response amplitude was gradually increased while the H-reflex amplitude was gradually decreased . Two consecutive recording will be taken and the mean H/M ratio will be calculated.

C. Musculoskeletal ultrasound assessment:

Sonographic evaluation will be performed using a linear transducer scanning frequency of ( 4-13 MHz) SAMSUNG MEDISON ( UGEO H 60) on the affected spastic calf muscles to qualify muscle echo intensity using the Heckmatt scale.

Radial extracorporeal shock wave therapy (r ESWT ) protocol:

Radial extracorporeal shock wave therapy (r ESWT) will be applied by Dornier AR2 machine (Dornier MedTech GmbH, Wessling, Germany) under ultrasound guidance, at musculotendinous junction of medial and lateral head of the gastrocnemius for spastic calf (gastrocnemius muscle and the soleus) muscles . 1.500 pulses will be applied by an R20 probe with a focusing depth of 4cm.The intensity will be 0.10 mJ to 0.3mJ/mm2 (2.5 bar), with frequency 4 Hz every week for one month for the treatment group and without operating the machine for the sham group . No anesthetic or analgesic drugs will be administered to patients during the therapy session. Both groups will be put under the same physiotherapeutic program performed by the same well-trained physiatrist .

ELIGIBILITY:
Inclusion Criteria:

* Adult ischemic or hemorrhagic hemiplegic patients who exhibited signs of unilateral spastic equinus foot for at least 6 months before the enrollment in the study will be selected to reduce the confounding effect of natural recovery.

Exclusion Criteria:

* Patients with fixed contractures or deformities at the ankle, fractures, cognitive impairment, different types of neuropathies or myopathies, implanted pacemaker and prior /or planned treatment using antispastic medications (i.e intrathecal baclofen or Botox injection ) or chemo -denervation ( phenol or alcohol nerve blocks ) within the last 6 months preceding the study , will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in modified Ashworth scale (MAS) for spastic plantar flexor muscles | about 6 months
Improvement of Passive ankle dorsiflexion range of motion ( PADFM) . | about 6 months
Reduction in time required to walk 10 meters (10 MWT). | about 6 months
Reduction in H/M ratio. | about 6 months
Change in spastic calf muscles echogenicity on Heckmatt scale. | about 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta University, Tanta, Elgharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided